CLINICAL TRIAL: NCT04786977
Title: Development of a Physiologic Measure of Vincristine Induced Peripheral Neuropathy in Children and Adolescents
Brief Title: Physiologic Measure of VIPN
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Julia Finkel, Principal Investigator, Children's National Research Institute
Other Study IDs: Pro00015693
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VIPN Patients
  Interventions: Other: No Intervention, Observational Study
- Healthy Volunteers
  Interventions: Other: No Intervention, Observational Study

INTERVENTIONS:
Other: No Intervention, Observational Study — No Intervention

SUMMARY:
The purpose of this study is the development of a physiologic endpoint using a novel technology that would provide an objective, easy to use and more sensitive assessment of VIPN in children and adolescents. The ability to more easily detect and monitor VIPN, even before it is clinically evident, would facilitate optimizing the dosing of vincristine for maximal disease response while minimizing the risk of lifelong functional deficits affecting quality of life. This approach would also enable the development of specific therapies to minimize or eliminate the occurrence of VIPN in children and adolescents. This is a single site study that aims to develop a novel device to evaluate and characterize vincristine-induced neuropathic pain. The investigators will enroll patients with ALL following the Delayed Intensification (DI) phase of treatment. At each study visit, the investigators will evaluate the nPRD as well as the TNS-PV. The nPRD will inform the neuropathy index which will be used to compare to the TNS-PV. We anticipate a correlation between the two.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years of age at the start of the study, are receiving vincristine in DI (clinical study population) and are willing and able to provide informed consent or assent to study participation.

Exclusion Criteria:

* have eye pathology which precludes pupillometry, are hemodynamically unstable, or are pregnant.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 30 patients and 10 healthy volunteers will be enrolled for this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of neuropathy index in patients with VIPN | 1 Year
  The primary objective of this study is the characterization of the neuropathy index in VIPN patients in order to measure VIPN severity.

SECONDARY OUTCOMES:
Correlation of neuropathy index with the TNS-PV | 1 Year
  The secondary objective is the correlation between the TNS-PV and the neuropathy index.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States